CLINICAL TRIAL: NCT01826565
Title: Comparison of Two Insertion Technique of I-gel: Standard Versus 90-degree Rotation
Brief Title: Comparison of Two Insertion Technique of I-gel
Acronym: I-gel90
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HPPark
Record Dates: First submitted 2013-03-19; First posted 2013-04-08 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Prostate Cancer; Prostate Tumor; Bladder Cancer; Bladder Tumor
Keywords: success
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): i-gel will be inserted without rotation
- Rotation (Experimental): Rotational technique applied
  Interventions: Procedure: Rotational technique

INTERVENTIONS:
Procedure: Rotational technique — 90 degree rotation
  Other Names: 90 degree rotation technique
  Arms: Rotation

SUMMARY:
To evaluate the efficacy of rotational technique in the insertion of i-gel

DETAILED DESCRIPTION:
The i-gel is one of the 2nd generation supraglottic airways. The rotational technique is known to increase the success rate of insertion of other supraglottic airways. The investigators try to evaluate the efficacy of rotational technique in the insertion of i-gel.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for general anesthesia(transurethral resection of bladder tumor or transurethral resection of the prostate) using i-gelTM

Exclusion Criteria:

* History of recent postoperative sore throat
* History of difficult airway
* Mouth opening < 2.5 cm
* Emergency operation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The success rate of insertion | up to 30 min.
  check oropharyngeal leakage at pressure 12 cmH2O

SECONDARY OUTCOMES:
postoperative sore throat | up to 2 days
  severe/moderate/minimal/none

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyung Park, MD PhD, Principal Investigator — Seoul National University of Hospital; Hyun-Chang Kim, MD, Principal Investigator — Seoul National University of Hospital